CLINICAL TRIAL: NCT03015623
Title: A Multi-center, Randomized, Sham-controlled, Double-blind, Ascending-dose Study of Extracorporeal Mesenchymal Stromal Cell Therapy (SBI-101 Therapy) in Subjects With Acute Kidney Injury Receiving Continuous Renal Replacement Therapy
Brief Title: A Study of Cell Therapy for Subjects With Acute Kidney Injury Who Are Receiving Continuous Renal Replacement Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sentien Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBI-101-01
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Acute Kidney Injury
Keywords: Mesenchymal stromal cells; MSC; Stem cells; Mesenchymal stem cells
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose cohort (Experimental): SBI-101 device containing 250 million MSCs
  Interventions: Biological: SBI-101
- High dose cohort (Experimental): SBI-101 device containing 750 million MSCs
  Interventions: Biological: SBI-101
- Control (Sham Comparator): Sham device containing no MSCs
  Interventions: Device: Sham

INTERVENTIONS:
Biological: SBI-101 — SBI-101 is a biologic/device combination product that combines two components: allogeneic human mesenchymal stromal cells (MSCs) and an FDA-approved plasmapheresis device. SBI-101 is administered via integration into a Continuous Renal Replacement Therapy circuit and is designed to regulate inflammation and promote repair of injured tissue.
  Arms: High dose cohort; Low dose cohort
Device: Sham — The sham control is an FDA-approved plasmapheresis device, without MSCs, which is integrated into a Continuous Renal Replacement Therapy circuit.
  Arms: Control

SUMMARY:
The purpose of this study is to assess the safety and tolerability of the investigational product, SBI-101, in subjects with Acute Kidney Injury (AKI) who require continuous renal replacement therapy. SBI-101 is a biologic/device combination product designed to regulate inflammation and promote repair of injured tissue using allogeneic human mesenchymal stromal cells.

The study will be conducted in two cohorts, with an interim analysis performed in between the cohorts. In the first cohort, subjects will be randomized to receive one of two treatments - low dose SBI-101 or sham control. In the second cohort, subjects will be randomized to receive one of two treatments - high dose SBI-101 or sham control. SBI-101 or sham control will be integrated into the renal replacement circuit and subjects in both cohorts will be treated for up to 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* AKI, as determined by the Investigator based on his/her clinical judgment
* Able to tolerate indwelling intravascular access
* Has tolerated Continuous Renal Replacement Therapy for at least 12 hours prior to IP treatment
* Likely to require Continuous Renal Replacement Therapy for at least an additional 48 hours
* Ability to give informed consent

Exclusion Criteria:

* Female subjects who are pregnant, planning to become pregnant, or lactating
* Known end-stage liver disease
* Hepatorenal syndrome
* Acute glomerulonephritis (e.g. rapidly progressive glomerulonephritis; membranoproliferative glomerulonephritis; post-streptococcal glomerulonephritis); acute interstitial nephritis (e.g. toxin- or drug- induced interstitial nephritis) or hereditary renal disease (e.g. Alport's Syndrome; polycystic kidney disease)
* AKI due to post-renal outflow obstruction
* Acute or chronic vasculitis of any etiology
* At the time of randomization, clinical evidence (e.g. febrile) suggestive of an uncontrolled or inadequately treated systemic infection
* History of a chronic systemic infection of any etiology regardless of therapy
* Active malignancy(-ies) and/or receiving active treatment for a malignancy(-ies), with the exception of non-melanoma skin cancer
* Subjects, who in the opinion of the Investigator, are likely to require escalating doses of vasopressors to attain and/or maintain hemodynamic stability
* Systemic immunosuppressive therapy that has not been stabilized for greater than 4 months, or in the case of chronic corticosteroid therapy, a dose of >15 mg/day of prednisone or the equivalent within the past 30 days
* Organ failure affecting more than 2 non-renal organs
* Platelet count <25,000/uL or other serious hematological abnormalities that would place subject in imminent danger of death
* Any prior medical condition that, in the judgment of the Investigator, would prevent the subject from safely participating in and/or completing all study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as measured by incidence of IP-related serious adverse events | Outcomes out to Day 28 and Serious Adverse Events through Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Brian Miller, Study Chair — Sentien Biotechnologies, Inc.
Locations (1):
- Lehigh Valley Hospital, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swaminathan M, Kopyt N, Atta MG, Radhakrishnan J, Umanath K, Nguyen S, O'Rourke B, Allen A, Vaninov N, Tilles A, LaPointe E, Blair A, Gemmiti C, Miller B, Parekkadan B, Barcia RN. Pharmacological effects of ex vivo mesenchymal stem cell immunotherapy in patients with acute kidney injury and underlying systemic inflammation. Stem Cells Transl Med. 2021 Dec;10(12):1588-1601. doi: 10.1002/sctm.21-0043. Epub 2021 Sep 28. PMID 34581517